CLINICAL TRIAL: NCT01800721
Title: A Randomized Controlled Trial to Train Black MSM as Peer Health Educators for HIV Testing and Prevention
Brief Title: Social Networks and Prevention for HIV Care and Prevention
Acronym: SNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Carl Latkin, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01DA031030 (NIH); 1R01DA031030 (NIH)
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: HIV
Keywords: HIV; testing; Social Network; African American; MSM; Men who have sex with men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Condition SNAP (Experimental): Behavioral Intervention SNAP HIV training and peer outreach
  Participants learn skills for sexual health and peer outreach which includes talking with network members about HIV testing and prevention.
  Interventions: Behavioral: SNAP
- SNAP Control Condition (Active Comparator): SNAP Control
  Participants receive information on HIV/STDs as well as healthy eating and nutrition instruction.
  Interventions: Behavioral: SNAP Control

INTERVENTIONS:
Behavioral: SNAP — Behavioral: SNAP 7 group sessions, and 1 individual session
  Other Names: Peer Education Randomized Controlled Trial for Black MSM for VCT and Prevention
  Arms: Experimental Condition SNAP
Behavioral: SNAP Control — Behavioral: SNAP control 7 group sessions
  Arms: SNAP Control Condition

SUMMARY:
The present study includes a randomized clinical trial of a peer health education intervention and a 12-month longitudinal study. The sample will include Black Men who have Sex with Men (MSM) who will be randomized into an experimental or control condition and then asked to recruit peer and risk network members for HIV testing over a 3 month period. Some of the network members who are recruited for voluntary counseling and testing (VCT) will enroll into the longitudinal study for assessments only. Both index and network participants will be assessed at baseline, 6, and 12-months.

The specific aims of the proposed study are to:

1. Train Black MSM (index participants in the experimental condition) to conduct peer health education, to promote VCT and HIV risk reduction among social network members, and to recruit social network members for VCT.
2. Examine changes in HIV risk behaviors and VCT among index participants and their network members in the experimental intervention as compared to those in the control condition.
3. Examine mediating effects of social environments (networks, social norms) on HIV risk behaviors and VCT, among indexes and network members.
4. Examine mediating effects of individual level factors (substance use and depression) on HIV risk behaviors and VCT among indexes and network members.

DETAILED DESCRIPTION:
The primary objective of this funded research is to conduct a randomized controlled trial of an experimental behavioral intervention that will train African American men who have sex with men (AA MSM) to 1) conduct peer health education, 2) to promote HIV risk reduction among their social network members, 3) promote HIV voluntary counseling and testing (VCT) among their social network members and 4) recruit social network members for VCT. Index participants are African American/Black men who have sex with men (MSM) who are randomized to either a peer education intervention or comparison condition. After the baseline is complete, index participants refer social network members (i.e. network participants) to the research clinic for HIV antibody testing. In addition, a subset of network participants participate in the longitudinal portion of the study.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for indexes include: (a) sex with a male partner within the prior 90 days; (b) self-reported Black or African American race/ethnicity; (c) self-reported biological male sex at birth; (d) identify as male; (e) unprotected vaginal or anal sex within the prior 90 days; (f) age 18 or older; (g) willingness to attend intervention sessions; (h) willingness to discuss HIV prevention and encourage VCT among network members; (i) reside in Baltimore city or a surrounding counties; (j) not planning on moving from Baltimore city or a surrounding county within the next year; (k) not involved in a behavioral intervention for HIV prevention within the prior five years.

Eligibility for network members for receiving VCT: (a) Provide a study coupon to verify that they were referred by an index participant and (b) age 18 or older.

Eligibility criteria for network members enrolling in the longitudinal study: (a) age 18 or older; (b) recruited by index participant and engaged in VCT at our clinic; (c) was either a current sex partner of index (male or female)or a Black MSM peer (as operationalized as self-reported black or African American and reporting sex with a man in the prior 90 days) and (d) had one of the following risk behaviors in the prior 90 days: unprotected vaginal or anal sex, diagnosed STI, or had sex with 2 or more people.

Exclusion Criteria:

Exclusion criteria for indexes include being previously enrolled in the study as a network participant.

Exclusion criteria for network participants include being previously enrolled in the study as an index participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2011-07-30 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Sex Risk Behavior at 6 months | 6 months
  We will measures sex risk behavior by assessing the frequency of oral and anal sex; frequency and consistency of condom use; the number and types (e.g., main, casual, and exchange) of sex partners in the prior 90 days; and the gender, sexual preference, and HIV and drug use status of each partner.
Change from Baseline in Sex Risk Behavior at 12 months | 12months
  We will measures sex risk behavior by assessing the frequency of oral and anal sex; frequency and consistency of condom use; the number and types (e.g., main, casual, and exchange) of sex partners in the prior 90 days; and the gender, sexual preference, and HIV and drug use status of each partner.
Change from Baseline in HIV Testing Rates at 6 months | 6 months
Change from Baseline in HIV Testing Rates at 12 months | 12 months
Number of Network Members Recruited for HIV Testing | 3 Months

SECONDARY OUTCOMES:
Change from Baseline in Drug Use at 6 months | 6 months
  Type of drug (e.g. cocaine, heroin, prescription drugs)and frequency of drug use
Change from Baseline in Drug Use at 12 months | 12 months
  Type of drug (e.g. cocaine, heroin, prescription drugs)and frequency of drug use

CONTACTS AND LOCATIONS:
Overall Officials: Carl Latkin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided